CLINICAL TRIAL: NCT01152996
Title: A Phase 3, Long-Term, Open-Label, Flexible-Dose, Extension Study Evaluating the Safety and Tolerability of Lu AA21004 (15 and 20 mg) in Subjects With Major Depressive Disorder
Brief Title: Safety and Tolerability of Vortioxetine (LuAA21004) - Open Label Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LuAA21004_314; U1111-1115-4927 (Registry Identifier: WHO)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Results first posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-04

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; Melancholia; Paraphrenia; Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vortioxetine (Experimental): Vortioxetine 10 mg, capsules, orally, once daily for the first week of treatment; then vortioxetine up-titrated to 15 mg or 20 mg, capsules, orally, once daily for up to 51 weeks.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine tablets
  Other Names: LuAA21004

SUMMARY:
The purpose of this study is to determine the long-term safety and tolerability of vortioxetine, once daily (QD), in participants with major depressive disorder.

DETAILED DESCRIPTION:
Depression has been recognized as a chronic illness that imposes a significant burden on individuals, families and society. Major depressive disorder (MDD) is among the most important causes of disability worldwide, in both developing and developed countries. Major depressive disorder is reported to be the most common mood disorder, with a lifetime prevalence of about 15% and as high as 25% in women. Major depressive disorder is characterized by the presence of 1 or more major depressive episodes that presents with depressed mood, loss of interest or pleasure, disturbed sleep or appetite, low energy, feelings of guilt or low self-worth, and poor concentration.

This is a multicenter extension study designed to allow eligible patients who have completed short-term efficacy and safety studies LuAA21004_315 (NCT01153009), LuAA21004_316 (NCT01163266) and LuAA21004_317 (NCT01179516) to receive the 52-week treatment with vortioxetine in this open-label extension study. Participants are expected to return to the site for approximately 13 visits.

A safety follow-up call will be made 4 weeks after completion of the 52-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Has completed either study LuAA21004_315 ( NCT01153009), LuAA21004_316 (NCT01163266), or LuAA21004_317 (NCT01179516) immediately prior to enrollment in the extension study (ie, the baseline visit is the same visit as the Week 8 [Lu AA21004_317] or Week 10 [Lu AA21004_315 or Lu AA21004_316] assessment of the preceding protocol).
* Suffers from a recurrent major depressive episode) as the primary diagnosis according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria (classification code 296.3x) at entry into the prior study.
* Twelve-month continuation treatment with Lu AA21004 is indicated for the treatment of this participant according to the opinion of the investigator.
* Females of childbearing potential who are sexually active with a nonsterilized male partner agree to routinely use adequate contraception throughout the duration of the study.

Exclusion Criteria:

* Has Major Depressive Disorder for whom other psychiatric disorders (mania, bipolar disorder, schizophrenia, or any psychotic disorder) have been diagnosed during the prior study.
* In the investigator's clinical judgment, has a significant risk of suicide and/or a score of ≥5 points on item 10 (suicidal thoughts) of the Montgomery Åsberg Depression Rating Scale (MADRS).
* In the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any reason.
* Has a clinically significant moderate or severe ongoing adverse event related to study medication from the prior study.
* Has used/uses disallowed concomitant medication.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1075 (Actual)
Dates: Start 2010-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 143 investigative sites in the United States from 07 Sep 2010 to 31 May 2013.
Pre-assignment Details: Patients who completed Studies LuAA21004_315 (NCT01153009), LuAA21004_316 (NCT01163266), and LuAA21004_317 (NCT01179516) and were willing to continue, and judged by the investigator to benefit from a 52-week continuation treatment with Lu AA21004, were enrolled and received flexible doses of study drug, based on patient response and tolerability.
Period: Overall Study
Arm/Group | Vortioxetine
Started | 1075
Treated | 1073
Completed | 538
Not Completed | 537
Not completed — Withdrawal by Subject | 142
Not completed — Adverse Event | 115
Not completed — Lost to Follow-up | 112
Not completed — Lack of Efficacy | 68
Not completed — Noncompliance | 41
Not completed — Other | 36
Not completed — Protocol Violation | 22
Not completed — Elevated liver enzymes | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vortioxetine
Number analyzed (Participants) | 1075
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 790
  Male | 285
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (or White, including Hispanic) | 813
  Black/African American | 249
  Asian | 7
  American Indian/Alaska Native | 5
  Native Hawaiian/Other Pacific Islander | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 104
  Non-Hispanic and Non-Latino | 971
Weight [Mean (Standard Deviation); unit: kg)] | 88.77 (24.160)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.60 (8.061)
Height [Mean (Standard Deviation); unit: cm] | 167.44 (9.456)
Montgomery Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: scores on a scale] — MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (i.e., apparent sadness, reported sadness, inner tension, etc.) rated on a 7-point Likert scale from 0 (normal) to 6 (most abnormal) with a total score range from 0 to 60. Higher scores indicate greater severity of symptoms.
  scores on a scale | 20.0 (10.70)
Hamilton Anxiety Scale (HAM-A) total score [Mean (Standard Deviation); unit: scores on a scale] — HAM-A is a 14 item rating scale to quantify anxiety symptomatology severity (i.e., anxious mood, tension, fear, insomnia, etc.) rated on a 5-point scale from 0 (not present) to 4 (severe) with a total score range from 0 to 56. Higher scores indicate greater severity of symptoms.
  scores on a scale | 11.6 (6.65)
Clinical Global Impression - Severity scale (CGI-S) score [Mean (Standard Deviation); unit: scores on a scale] — The CGI-S assesses the clinician's impression of the subject's current state of mental illness and consists of one question for the investigator: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on a seven-point scale (1=normal, not ill at all; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill). Higher scores indicate greater severity of illness.
  scores on a scale | 3.3 (1.21)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events at a Frequency Threshold of ≥5%
Description: Treatment-emergent adverse events (TEAE) are adverse events with an onset that occurs after receiving study drug and within 30 days after receiving the last dose of study drug. A TEAE may also be a pretreatment adverse event or a concurrent medical condition diagnosed prior to the date of first dose of study drug that increases in severity after the start of dosing.
Time Frame: Over the 52 week period
Population: Safety set
Measure: Number; unit: participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 1073
participants
  Nausea | 258
  Diarrhea | 80
  Vomiting | 68
  Constipation | 65
  Nasopharyngitis | 68
  Viral upper respiratory tract infection | 66
  Upper respiratory tract infection | 60
  Weight increased | 65
  Headache | 136
  Insomnia | 56

2. Primary Outcome: Number of Participants With Serious Treatment-Emergent Adverse Events
Description: Serious treatment-emergent adverse events (serious-TEAE) are adverse events with an onset that occurs after receiving study drug and within 30 days after receiving the last dose of study drug. A serious-TEAE may also be a pretreatment adverse event or a concurrent medical condition diagnosed prior to the date of first dose of study drug that increases in severity after the start of dosing. Serious Adverse Events include adverse events that result in death, require either inpatient hospitalization or the prolongation of hospitalization, are life-threatening, result in a persistent or significant disability/incapacity or result in a congenital anomaly/birth defect. Other important medical events, based upon appropriate medical judgment, may also be considered serious adverse events if a trial participant's health is at risk and intervention is required to prevent an outcome mentioned.
Time Frame: Over the 52 week period
Population: Safety set
Measure: Number; unit: participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 1073
participants | 29

3. Primary Outcome: Treatment-Emergent Adverse Events Leading to Study Discontinuation
Description: Treatment-emergent adverse events are adverse events with an onset that occurs after receiving study drug and within 30 days after receiving the last dose of study drug. A TEAE may also be a pre-treatment adverse event or a concurrent medical condition diagnosed prior to the date of first dose of study drug that increases in severity after the start of dosing.
Time Frame: Over the 52 week period
Population: Safety set
Measure: Number; unit: participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 1073
participants | 117

4. Secondary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The change between MADRS total score at each assessed visit and MADRS score at baseline. MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (i.e., apparent sadness, reported sadness, inner tension, etc.) rated on a 7-point Likert scale from 0 (normal) to 6 (most abnormal) with a total score range from 0 to 60. Higher scores indicate greater severity of symptoms.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 36, 44, and 52
Population: Safety set, observed cases (OC)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 1043
units on a scale
  Week 1 (n=1043) | -2.7 (6.32)
  Week 2 (n=1043) | -4.8 (7.50)
  Week 4 (n=1004) | -6.1 (8.50)
  Week 8 (n=936) | -7.9 (9.19)
  Week 12 (n=843) | -8.5 (9.55)
  Week 16 (n=777) | -9.1 (9.50)
  Week 20 (n=747) | -9.4 (10.03)
  Week 24 (n=697) | -9.7 (9.64)
  Week 28 (n=670) | -9.5 (10.20)
  Week 36 (n=617) | -9.7 (10.44)
  Week 44 (n=573) | -10.3 (10.70)
  Week 52 (n=534) | -10.3 (11.00)

5. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score
Description: The change between HAM-A score at each assessed visit and HAM-A score at baseline. HAM-A is a 14 item rating scale to quantify anxiety symptomatology severity (i.e., anxious mood, tension, fear, insomnia, etc.) rated on a 5-point scale from 0 (not present) to 4 (severe) with a total score range from 0 to 56. Higher scores indicate greater severity of symptoms.
Time Frame: Baseline and Weeks 4, 24, and 52
Population: Safety set, observed cases (OC)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 1029
units on a scale
  Week 4 (n=1029) | -2.6 (4.98)
  Week 24 (n=742) | -4.2 (5.84)
  Week 52 (n=548) | -4.8 (6.52)

6. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale-Severity of Illness (CGI-S)
Description: The change between CGI-S score at each assessed visit and CGI-S score at baseline. The CGI-S assesses the clinician's impression of the subject's current state of mental illness and consists of one question for the investigator: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on a seven-point scale (1=normal, not ill at all; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=extremely ill). Higher scores indicate greater severity of illness.
Time Frame: Baseline and Weeks 4, 24, and 52
Population: Safety set, observed cases (OC)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 1030
units on a scale
  Week 4 (n=1030) | -0.6 (0.99)
  Week 24 (n=743) | -1.0 (1.16)
  Week 52 (n=549) | -1.2 (1.32)

7. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score
Description: The change between the SDS total score at each assessed visit and the total score collected at baseline. The SDS is a 3 item rating scale to assess functional impairment (panic, anxiety, phobic and depressive symptoms) over three inter-related domains (work/school, social life, and family life/home responsibilities) rated on an 11 point scale from 0 (not at all) to 10 (extremely) with a total score range from 0 to 30. Higher scores indicate greater severity of impairment.
Time Frame: Baseline and Weeks 12, 24, 36, and 52
Population: Safety set, observed cases (OC)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 650
units on a scale
  Week 12 (n=650) | -2.8 (6.69)
  Week 24 (n=494) | -3.9 (6.88)
  Week 36 (n=414) | -4.0 (7.37)
  Week 52 (n=381) | -4.7 (7.11)

8. Secondary Outcome: Change From Baseline in SDS Work/School Subscale
Description: The change between the Sheehan Disability work/school subscale score at each assessed visit and work/school subscale score collected at baseline. The SDS is a 3 item rating scale to assess functional impairment (panic, anxiety, phobic and depressive symptoms) over three inter-related domains (work/school, social life, and family life/home responsibilities) rated on an 11 point scale from 0 (not at all) to 10 (extremely). Higher scores indicate greater severity of impairment.
Time Frame: Baseline and Weeks 12, 24, 36, and 52
Population: Safety set, observed cases (OC)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 650
units on a scale
  Week 12 (n=650) | -0.8 (2.42)
  Week 24 (n=494) | -1.2 (2.48)
  Week 36 (n=414) | -1.2 (2.60)
  Week 52 (n=381) | -1.4 (2.61)

9. Secondary Outcome: Change From Baseline in SDS Social Life Subscale
Description: The change between the Sheehan Disability social life subscale score at each assessed visit and social life subscale score collected at baseline. The SDS is a 3 item rating scale to assess functional impairment (panic, anxiety, phobic and depressive symptoms) over three inter-related domains (work/school, social life, and family life/home responsibilities) rated on an 11 point scale from 0 (not at all) to 10 (extremely). Higher scores indicate greater severity of impairment.
Time Frame: Baseline and Weeks 12, 24, 36, and 52
Population: Safety set, observed cases (OC)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 942
units on a scale
  Week 12 (n=942) | -1.0 (2.53)
  Week 24 (n=721) | -1.4 (2.55)
  Week 36 (n=617) | -1.4 (2.82)
  Week 52 (n=545) | -1.6 (2.85)

10. Secondary Outcome: Change From Baseline in SDS Family Life/Home Responsibilities Subscale
Description: The change between the Sheehan Disability family life/home responsibilities subscale score at each assessed visit and family life/home responsibilities subscale score collected at baseline. The SDS is a 3 item rating scale to assess functional impairment (panic, anxiety, phobic and depressive symptoms) over three inter-related domains (work/school, social life, and family life/home responsibilities) rated on an 11 point scale from 0 (not at all) to 10 (extremely). Higher scores indicate greater severity of impairment.
Time Frame: Baseline and Weeks 12, 24, 36, and 52
Population: Safety set, observed cases (OC)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 942
units on a scale
  Week 12 (n=942) | -0.9 (2.39)
  Week 24 (n=721) | -1.3 (2.47)
  Week 36 (n=617) | -1.4 (2.74)
  Week 52 (n=545) | -1.6 (2.76)

ADVERSE EVENTS:
Time Frame: 56 weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vortioxetine
Serious Adverse Events (participants affected / at risk) | 29/1073
Other Adverse Events (participants affected / at risk) | 854/1073
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=1073)
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Esophageal rupture (Gastrointestinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Anal abscess (Infections and infestations) | 1
Latent syphilis (Infections and infestations) | 1
Periorbital cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Wound sepsis (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Complicated migraine (Nervous system disorders) | 1
Transient ischemic attack (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Suicide attempt (Psychiatric disorders) | 3
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Phlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=1073)
Nausea (Gastrointestinal disorders) | 258
Diarrhea (Gastrointestinal disorders) | 80
Vomiting (Gastrointestinal disorders) | 68
Constipation (Gastrointestinal disorders) | 65
Nasopharyngitis (Infections and infestations) | 68
Viral upper respiratory tract infection (Infections and infestations) | 66
Upper respiratory tract infection (Infections and infestations) | 60
Weight increased (Investigations) | 65
Headache (Nervous system disorders) | 136
Insomnia (Nervous system disorders) | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.